CLINICAL TRIAL: NCT00790361
Title: Mapping the Natural History of Traumatic Spinal Cord Injury in the Sensorimotor Cortex Using Functional Magnetic Resonance Imaging, Magnetic Resonance Spectroscopy and Diffusion Tensor Imaging
Brief Title: The Natural History of Traumatic Spinal Cord Injury Using fMRI, MRS and DTI
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 13652
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Central Cord Syndrome
Keywords: cervical spondylotic myelopathy; spinal cord compression; magnetic resonance spectroscopy; functional magnetic resonance imaging; brain plasticity
MeSH Terms: conditions — Central Cord Syndrome; Spinal Cord Compression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Controls (healthy volunteers) will have two scans (fMRI, MRS and DTI) six months apart to determine reproducibility.
  A blinded investigator will administer JOA, ASIA/ISCOS, NDI and SF-36 prior to the scan at all time points.
- CCS Participants: CCS participants will have three scans (fMRI, MRS and DTI), one acutely (up to 48 hours after injury), one subacutely (15 days after injury), and one late (6 months after injury).
  A blinded investigator will administer JOA, ASIA/ISCOS, NDI and SF-36 prior to the scan at all time points.

SUMMARY:
Traumatic spinal cord injury is a common injury to the spine and can lead to a clinical syndrome called central cord syndrome (CCS). CCS is an incomplete spinal cord injury where one starts to lose more motor function in the upper rather than lower extremities. It affects a wide range of the population from the young to the old. However, the natural history of CCS is poorly understood.

Research has shown that the injury resulting in CCS might be due to the pinching or compressing of the spinal cord. This creates damage to a part of the spinal cord and creates difficulties in the signal getting through. We believe that we can gain a better understanding of the natural history of incomplete spinal cord injury as well as the recovery process.

It is possible to track many changes in the brain and motor function through a variety of methods. One can track the concentrations of different chemicals (metabolites) by using magnetic resonance spectroscopy (MRS), changes in brain activation by using functional magnetic resonance imaging (fMRI) and thread-like nerve fibers in the spine by using diffusion tensor imaging (DTI). In our study we will be detecting differences in brain metabolism and activation of different parts of the brain during specific movement and in the nerve fibers in the brain.

We hypothesize that there will be decreased levels of N-acetylaspartate (NAA, a putative marker of neuronal function) and decreased levels of glutamate (the primary excitatory neurotransmitter) in the motor cortex in patients with CCS when compared with controls. Over time, we hypothesize that the normalization of metabolite levels will correlate with the extent of neurologic recovery. We also hypothesize a reorganization of brain activation patterns with time such that patients will show increased volumes of activation in the motor cortex with recovery and that this will correlate with the extent of neurologic outcome. Over time, we predict that there will be normalization of the fibre track anatomy that will correlate with neurological recovery.

DETAILED DESCRIPTION:
The long-term goal of this project is to develop predictors of neurological recovery based on brain metabolism, brain activation patterns, and fibre tracks in patients with traumatic CCS. The objective of this preliminary study is to evaluate metabolic changes, brain activation pattern reorganization and altered spinal cord fibre tracks in patients suffering from traumatic CCS to gain a better understanding of the natural history of this condition. Magnetic resonance spectroscopy (MRS), functional magnetic resonance imaging (fMRI), and diffusion tensor imaging (DTI) will be used to investigate the changes in brain metabolite concentrations, cerebral cortical activation, and fibre tract anatomy, respectively, in patients and controls.

Ten patients having traumatic CCS will be recruited from the Clinical Neurological Sciences Department at the London Health Sciences Centre, University Campus. All participants will undergo an fMRI, MRS and DTI scan of the motor cortex to measure the volume of activation, signal intensity and levels of NAA and glutamate. The CCS participants will have three scans, one acutely (up to 48 hours after injury), one subacutely (15 days after injury), and one late (6 months after injury). Healthy volunteers will have two scans six months apart to determine reproducibility.

Clinical changes will be measured using validated disease specific scoring instruments including the Japanese Orthopedic Association scale (JOA), ASIA/ISCOS Impairment Scale, and the Neck Disability Index (NDI). General quality of life will be measured using the 36-item Short-Form Health Survey (SF-36). A blinded investigator will administer these instruments prior to the scan at all time points.

ELIGIBILITY:
Inclusion Criteria:

* between 30 and 85 years of age
* right handed
* with normal/corrected hearing and vision
* fluent in reading and speaking Canadian or American English
* able to follow simple task instructions
* able to maintain standardized movements
* available to return for the 15 day and 6 month imaging sessions
* competent to give consent

Exclusion Criteria:

* must not have any other neurological disorder or systemic disease that may affect neurologic function
* not have any potential magnetic metal fragments in their body
* suffering from claustrophobia
* having a pacemaker or other electronic implants
* have been or currently is a welder or soldier
* have been injured by a metallic object that has not been removed
* pregnant or trying to conceive
* have cerebral aneurysm clips

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ten patients and ten controls will be recruited from the Clinical Neurological Sciences outpatient clinic at the London Health Sciences Centre, University Campus
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-06-18 (Actual); Primary Completion 2010-01-31 (Actual); Study Completion 2010-01-31 (Actual)

PRIMARY OUTCOMES:
Measure the volume of activation, signal intensity and levels of NAA and glutamate using fMRI, MRS and DTI. | acutely (up to 48 hours after injury), subacutely (15 days after injury), and late (6 months after injury)

SECONDARY OUTCOMES:
Clinical changes will be measured using validated disease specific scoring instruments including the Japanese Orthopedic Association scale (JOA), ASIA/ISCOS Impairment Scale, and the Neck Disability Index (NDI). | Acutely (up to 48 hours after injury), subacutely (15 days after injury), and late (6 months after injury)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Duggal, M.D., MSc, Principal Investigator — London Health Research Institute, London Health Sciences Centre
Locations (1):
- London Health Sciences Center, University Campus, London, Ontario, Canada

REFERENCES:
- [Background] Aito S, D'Andrea M, Werhagen L, Farsetti L, Cappelli S, Bandini B, Di Donna V. Neurological and functional outcome in traumatic central cord syndrome. Spinal Cord. 2007 Apr;45(4):292-7. doi: 10.1038/sj.sc.3101944. Epub 2006 Jun 13. PMID 16773038
- [Background] Clark CA, Werring DJ. Diffusion tensor imaging in spinal cord: methods and applications - a review. NMR Biomed. 2002 Nov-Dec;15(7-8):578-86. doi: 10.1002/nbm.788. PMID 12489104
- [Background] De Stefano N, Matthews PM, Arnold DL. Reversible decreases in N-acetylaspartate after acute brain injury. Magn Reson Med. 1995 Nov;34(5):721-7. doi: 10.1002/mrm.1910340511. PMID 8544693
- [Background] Dvorak MF, Fisher CG, Hoekema J, Boyd M, Noonan V, Wing PC, Kwon BK. Factors predicting motor recovery and functional outcome after traumatic central cord syndrome: a long-term follow-up. Spine (Phila Pa 1976). 2005 Oct 15;30(20):2303-11. doi: 10.1097/01.brs.0000182304.35949.11. PMID 16227894
- [Background] Holly LT, Dong Y, Albistegui-DuBois R, Marehbian J, Dobkin B. Cortical reorganization in patients with cervical spondylotic myelopathy. J Neurosurg Spine. 2007 Jun;6(6):544-51. doi: 10.3171/spi.2007.6.6.5. PMID 17561743
- [Background] Kassem MN, Bartha R. Quantitative proton short-echo-time LASER spectroscopy of normal human white matter and hippocampus at 4 Tesla incorporating macromolecule subtraction. Magn Reson Med. 2003 May;49(5):918-27. doi: 10.1002/mrm.10443. PMID 12704775
- [Background] Pickett GE, Campos-Benitez M, Keller JL, Duggal N. Epidemiology of traumatic spinal cord injury in Canada. Spine (Phila Pa 1976). 2006 Apr 1;31(7):799-805. doi: 10.1097/01.brs.0000207258.80129.03. PMID 16582854
- [Background] Puri BK, Smith HC, Cox IJ, Sargentoni J, Savic G, Maskill DW, Frankel HL, Ellaway PH, Davey NJ. The human motor cortex after incomplete spinal cord injury: an investigation using proton magnetic resonance spectroscopy. J Neurol Neurosurg Psychiatry. 1998 Nov;65(5):748-54. doi: 10.1136/jnnp.65.5.748. PMID 9810950
- [Background] Yamazaki T, Yanaka K, Fujita K, Kamezaki T, Uemura K, Nose T. Traumatic central cord syndrome: analysis of factors affecting the outcome. Surg Neurol. 2005 Feb;63(2):95-9; discussion 99-100. doi: 10.1016/j.surneu.2004.03.020. PMID 15680638